CLINICAL TRIAL: NCT04813393
Title: Psychometric Properties of Compliance of Parents of Children With Cerebral Palsy to Home Program Questionnaire
Brief Title: Compliance of Parents of Children With Cerebral Palsy to Home Program Questionnaire
Acronym: CoPoCPHP
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Mintaze Kerem Gunel, Prof. Doc.Dr., Hacettepe University
Other Study IDs: GO: 20/357
Record Dates: First submitted 2021-03-21; First posted 2021-03-24 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Cerebral Palsy
Keywords: home program; cerebral palsy; questionnaire development; parent
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Compliance of Parents of Children with Cerebral Palsy to Home Program Assesment Questionnaire Group: The CPHP-Q was administered as a caregiver-report questionnaire. It aims to measure home program adherence of parents of children with CP. Parents applied this instrument in the study.
  Interventions: Other: Questionnaire Development

INTERVENTIONS:
Other: Questionnaire Development — To evaluate psychometric the properties of the Compliance of Parents of Children with Cerebral Palsy to Home Program Assesment Questionnaire (CPHP-Q), a caregiver-report for adherence and frequency of home program implementation of parents of children with Cerebral Palsy.

SUMMARY:
This study aims to evaluate the psychometric properties of the Compliance of Parents of Children with Cerebral Palsy to Home Program Assesment Questionnaire (CPHP-Q), a caregiver-report for adherence and frequency of home program implementation of parents of children with Cerebral Palsy.

ELIGIBILITY:
Inclusion Criteria:

1. having a child with CP 2 to 18 years,
2. being a primary caregiver,
3. understanding of Turkish without an interpreter, and Turkish literacy,

Exclusion Criteria:

1. having any chronic illness or disability to prevent the home program,
2. haven't applied home program before.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Participants in the current study were parents of chlidren with 2 to 18 years and recruited at Hecettepe Univercity Physical Therapy and Rehabilitation Faculty Cerebral Palsy and Pediatric Rehabilitation Unit.
Sampling Method: Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Compliance of Parents of Children with Cerebral Palsy to Home Program Assesment Questionnaire (CPHP-Q) | At baseline
  The CPHP-Q was administered as a caregiver-report questionnaire. It aims to measure home program adherence of parents of children with CP. İt consist of 22 items. The highest score 110, the lowest score 22.

SECONDARY OUTCOMES:
Assessment of Life Habits for Children questionnaire (LIFE-H) | At baseline
  The questionnaire was designed and validated to assess the social participation of children with disabilities. It consists of 11 category: nutrition, physical fitness, personal care, mobility, interpersonal communication, social roles, education, recreational activities, responsibilities, housing, and social life. Each Life-H item is ranked on a 0 to 9 scale for accomplishment, where a score of 0 represents "not accomplished" and a score of 9 equals "no difficulty and no assistance."

CONTACTS AND LOCATIONS:
Overall Officials: Mutlu Hayran, PhD, Study Chair — Hacettepe Univercity; Meltem Şengelen, PhD, Study Chair — Hacettepe Univercity
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No